CLINICAL TRIAL: NCT04923256
Title: AAT-APP+: A Pilot RCT of a Novel Smart-phone App to Reduce Alcohol Consumption Among Middle to Older Adults in the Eastern Health Community
Brief Title: AAT-APP+: A Novel Brain-training App to Reduce Drinking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turning Point (Other)
Collaborators: Monash University (Other); Eastern Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 73140
Record Dates: First submitted 2021-05-11; First posted 2021-06-11 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2022-07

CONDITIONS: Alcohol Use Disorder
Keywords: Alcohol; Intervention; Cognitive Bias Modification; Mobile Health Intervention; Approach Bias
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blinded (Participant, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Approach Bias Modification (Experimental): Participants will complete 2 x 5-7 min training sessions of approach bias modification for the period of four weeks
  Interventions: Behavioral: AAT-APP: A novel smart-phone approach-avoidance bias modification intervention
- Control: Minimal intervention (Active Comparator): Participants will complete a standardised alcohol approach-avoidance training task (AAT) on a weekly basis for four weeks.
  Interventions: Behavioral: Sham training control

INTERVENTIONS:
Behavioral: AAT-APP: A novel smart-phone approach-avoidance bias modification intervention — Participants allocated to the intervention group will be required to upload photos of drinks they wish to avoid, as well as activities they wish to engage in more, and be trained to avoid and approach by repeatedly 'swiping' images away from and towards themselves, respectively.
  Arms: Experimental: Approach Bias Modification
Behavioral: Sham training control — Complete an AAT on a weekly basis for four weeks
  Arms: Control: Minimal intervention

SUMMARY:
This study will explore the feasibility, acceptability, and preliminary effectiveness of a smart phone delivered form of cognitive training intervention (Approach Bias Modification (ABM)) in a non-clinical community sample of middle to older adults (>55 years) reporting hazardous alcohol use in a pilot randomised controlled trial (RCT). This app is called AAT-APP+

DETAILED DESCRIPTION:
Alcohol use in older adults is of particular concern, with the 55-74 year old cohort most likely to exceed lifetime alcohol risk. Approach Bias Modification (ABM) is a form of computerised cognitive training that is an efficacious intervention for alcohol use disorder. Previous studies are limited in that the stimuli are not personalised, nor are interventions readily accessible to non-treatment seeking problem drinkers. This has led to the development of a world-first, smart phone version of ABM called AAT-APP+

The current study aims to explore the feasibility, acceptability, and preliminary effectiveness of AAT-APP+ in reducing alcohol consumption and cravings in a pilot RCT with a non-clinical community sample of 100 older adults (aged 55+ years) reporting hazardous alcohol use (i.e. a score of 8+ on the AUDIT), recruited via targeted advertising. Participants in active training will upload (or select pre-selected) photos of beverages and meaningful activities, which will form the 'avoid' and 'approach' stimuli, respectively, then complete two training sessions per week for four weeks, with results compared to controls. AAT-APP+ holds promise as an innovate, cost-effective, and remotely accessible adjunctive support tool.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 55+ years
* Score 8 or higher on the Alcohol Use Disorders Identification Test (indicates 'hazardous' levels of alcohol use).
* Access to an Android or Apple smart phone and Australian contact number
* Wish to reduce their drinking
* Live within the Eastern Health Primary and Secondary Catchment (see map below)

Exclusion Criteria:

* Under age 55
* Not concerned about their drinking
* Do not wish to reduce their alcohol use in the next 4-6 weeks
* Do not reside with the appropriate catchment will be excluded.
* Experiencing severe alcohol problems likely to need professional treatment (i.e. presence of withdrawal symptoms in the past year)

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Change in number of standard drinks past week | Change from baseline standard drinks at 4-weeks
  Change from baseline in number of standard drinks at 4-weeks

SECONDARY OUTCOMES:
Change in number of drinking days past week | Change from baseline drinking days at 4-weeks
  Change from baseline in number of drinking days at 4-weeks
Change in number of standard drinks consumed in the past week throughout the 4-week training program | Change from baseline standard drinks consumed in the week prior to training compared to each week of training (i.e. week 1, week 2, week 3).
  Change from baseline in number of standard drinks at the end of each week of training (i.e. week 1, week 2, week 3)
Change in number of drinking days past week throughout the 4-week training program | Change from baseline number of drinking days in the week prior to training compared to each week of training (i.e. week 1, week 2, week 3).
  Change from baseline in the number of drinking days at the end of each week of training (i.e. week 1, week 2, week 3)
Change in number of drinking days at follow up | Change from baseline number of drinking days at 8-weeks
  Change from baseline in the number of drinking days at 8-weeks
Craving Frequency Score (as measured by the Craving Experience Questionnaire, Frequency) | Change from baseline craving frequency at 4-weeks
  Change from baseline craving, as measured by the Craving Experience Questionnaire, at 4-weeks. The Craving Experience Questionnaire - frequency consists of an 11-point visual analogue scale, anchored 0 = not at all, to 10 = extremely/constantly, assessing craving frequency, whereby higher scores are suggestive of greater craving frequency
Craving Frequency Score (as measured by the Craving Experience Questionnaire, Frequency, Follow up) | Change from baseline craving frequency at 8-weeks
  Change from baseline craving, as measured by the Craving Experience Questionnaire, at 8-weeks. The Craving Experience Questionnaire - frequency consists of an 11-point visual analogue scale, anchored 0 = not at all, to 10 = extremely/constantly, assessing craving frequency, whereby higher scores are suggestive of greater craving frequency
Approach-avoidance behaviours (alcohol approach avoidance questionnaire) | Change from baseline approach-avoidance behaviours at 4-weeks
  Change from baseline in self-report of approach and avoidance towards alcohol, as measured by the alcohol approach avoidance questionnaire, at 4-weeks. This is a 20-item self report measure with two primary dimensions of alcohol craving (i.e. approach and avoidance), where higher scores are suggestive of greater approach or avoidance behaviours (rated on a 9-point scale, 0 = not at all, 8 = very strongly).
Approach-avoidance behaviours (alcohol approach avoidance questionnaire) at follow up | Change from baseline approach-avoidance behaviours at 8-weeks
  Change from baseline in self-report of approach and avoidance towards alcohol, as measured by the alcohol approach avoidance questionnaire, at 8-weeks. This is a 20-item self report measure with two primary dimensions of alcohol craving (i.e. approach and avoidance), where higher scores are suggestive of greater approach or avoidance behaviours (rated on a 9-point scale, 0 = not at all, 8 = very strongly).
Approach-avoidance behaviours (approach avoidance task) | Change in alcohol approach/avoidance from baseline at 4-weeks
  Change in alcohol approach/avoidance behaviours from baseline at 4-weeks, as calculated by([reaction time for pushing alcohol stimuli] - [reaction time for pulling alcohol related stimuli]) - ([reaction time for pushing neutral objects] - [reaction time for pulling neutral objects]). Higher positive values indicate a tendency to approach alcohol faster (i.e. faster reaction times for pulling as opposed to pushing), whereas negative values indicate a tendency to avoid alcohol (i.e. slower reactions times for pulling compared to pushing alcohol).
Change in quality of life, as measured by the Australian Treatment Outcomes Profile Questionnaire | Change in quality of life from baseline at 4-weeks
  Change in self report of quality of life from baseline, as measured by the quality of life items from the Australian Treatment Outcomes Profile, at 4-weeks. This is a score ranging from 0-10, whereby higher scores are indicative of greater quality of life.
Change in quality of life, as measured by the Australian Treatment Outcomes Profile Questionnaire at follow up | Change in quality of life from baseline at 8-weeks
  Change in self report of quality of life from baseline, as measured by the quality of life items from the Australian Treatment Outcomes Profile, at 8-weeks. This is a score ranging from 0-10, whereby higher scores are indicative of greater quality of life.
Change in subjective cognitive concerns | Change from baseline in subjective cognitive concerns at 4-weeks
  Change from baseline in subjective ratings of cognitive concerns, as measured by responses to the question "How concerned are you about changes in your thinking, attention, or memory skills", at 4 weeks. Participants will respond on a 5-point visual analogue scale ranging from 0 = not at all to 5 = extremely concerned, whereby higher scores indicate a greater degree of concern in relation to cognition
Change in subjective cognitive concerns at follow up | Change from baseline in subjective cognitive concerns at 8-weeks
  Change from baseline in subjective ratings of cognitive concerns, as measured by responses to the question "How concerned are you about changes in your thinking, attention, or memory skills", at 8 weeks. Participants will respond on a 5-point visual analogue scale ranging from 0 = not at all to 5 = extremely concerned, whereby higher scores indicate a greater degree of concern in relation to cognition
Change in number of standard drinks at follow up | Change from baseline in number of drinking days at 8 weeks
  Change from baseline in number of drinking days at 8 weeks
Change in severity of alcohol dependence, as measured by the Severity of Dependence Scale | Change in severity of alcohol dependence at 4-weeks
  Change from baseline in severity of alcohol dependence, as measured by the Severity of Dependence Scale, at 4 weeks. Participants respond to five items on a 4-point scale (each scored from 0-3), with total scores ranging from 0-15 where higher scores indicate greater severity of alcohol dependence.
Change in severity of alcohol dependence (SDS) at follow up | Change in severity of alcohol dependence at 8-weeks
  Change from baseline in severity of alcohol dependence, as measured by the Severity of Dependence Scale, at 8-weeks. Participants respond to five items on a 4-point scale (each scored from 0-3), with total scores ranging from 0-15 where higher scores indicate greater severity of alcohol dependence.

OTHER OUTCOMES:
Task acceptability as measured by the Mobile Application Rating Scale - user version (uMARS) | 4-weeks
  Acceptability of the SWIPE app, as measured by the user version of the Mobile Application Rating Scale (uMARS). Participants will respond on a scale of 1-5, whereby higher scores indicate greater acceptability
Task feasibility | 4-weeks
  Feasibility of SWIPE app, as measured by recruitment and completion rates of at least 100 older adults within 6-months of advertising, with 50% of participants completing at least four sessions

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Manning, PhD, Principal Investigator — Turning Point
Locations (1):
- Turning Point, Richmond, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No
A layman summary of the research findings will be made available on the Turning Point website. Participants are told in the explanatory statement that if they would like to be informed of the research findings directly, they will need to contact the researchers via email. Should participants request results of research, this will be in aggregate form.